CLINICAL TRIAL: NCT03425266
Title: Incorporating Patient Preferences Into Decisions About Chronic Pain Management (The Pain APP Study)
Brief Title: The Pain App Study: A Novel Shared Decision Making Tool for People With Chronic Pain
Acronym: PainApp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shared Decision Making Resources (Other)
Collaborators: University of New England (Other); Pfizer (Industry)
Responsible Party: Principal Investigator, Nananda Col, Principal Investigator, Shared Decision Making Resources
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 012616-019
Record Dates: First submitted 2018-01-12; First posted 2018-02-07 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Chronic Pain
Keywords: shared decision-making; decision support tool; patient-provider communication; managing chronic pain; patient preferences; values clarification
MeSH Terms: conditions — Chronic Pain; Patient Preference

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either the new intervention (PainApp) or a website designed for people with chronic pain before an upcoming appointment with their provider.
Who Masked: Participant, Care Provider
Masking Description: Participants are not aware of whether they are in the treatment or control group. Providers are not informed which group a patient is in, however, because the intervention generates a summary page that the patient may choose to send to their provider, the provider would be aware of a patients' group assignment if they shared the summary with the provider.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive decision support tool (Experimental): Online interactive multimedia decision support tool that the patient interacts with before seeing their provider that helps them learn more about chronic pain, identify treatment goals and preferences, and communicate more effectively with their provider. The tool takes between 20-45 minutes to use. It generates and transmits a preference summary for the patient and a summary of relevant shared decision making elements and medical history elements intended for sharing with providers if the patient chooses.
  Interventions: Other: Interactive decision support tool
- Control (No Intervention): Our control arm is a leading consumer-facing website designed for people with chronic pain (the ACPA). Subjects randomly assigned to this arm will be directed to the page focusing on communication tools, which also includes links to other parts of the website. The specific page is: https://theacpa.org/Communication-Tools

INTERVENTIONS:
Other: Interactive decision support tool — PainApp 1) assesses patient treatment goals (a structured values clarification exercise) and preferences, including decision making and communication preferences; 2) presents structured educational modules tailored to the user's stated goals and preferences; 3) presents educational information addressing identified gaps in care and communication; 4) assesses pain, pain interference, function, and other clinical factors; 5) generates succinct individualized summaries of patient treatment preferences and medical history, tailored to different clinical settings; 6) generates a personalized report for the patient, based on their goals and interests; 7) transmits the clinical summary to the patient and their provider(s), with patient permission.
  Other Names: PainApp
  Arms: Interactive decision support tool

SUMMARY:
The investigators seek to understand the preferences, goals, and perspectives of patients with chronic pain and their health care providers (HCPs) to create a patient-centered decision support tool. This tool, aimed at patients and HCPs, should improve patient-provider communication and chronic pain management. The investigators' long-term goal is to improve the quality of life of patients with chronic pain. The investigators target adults with chronic unremitting pain and HCPs who manage patients with chronic pain, including primary care providers and pain specialists.

A pilot randomized controlled trial (RCT) will measure the impact of a new online tool that the investigators developed (Pain-APP) in a representative sample of adults with chronic pain, including approximately 50 patients and 4-15 HCPs. Eligible patients will be enrolled online, and after informed consent and eliciting baseline socio-demographic information, randomized online to either Pain-APP or the control group, which will consist of online educational materials at the ACPA website (https://theacpa.org/Communication-Tools). Patients in both groups will be assessed online before, just after viewing the intervention materials, just after the index clinic visit, and 1 month later. Patient-reported outcomes include patient-provider communication, pain intensity and interference, attitudes towards and use of opioid medication.

DETAILED DESCRIPTION:
Having completed our formative work, development and refinement of PainApp, the investigators will evaluate it in a small pilot randomized controlled trial (RCT) on a representative sample of patients with chronic pain and their HCPs.

The investigators will conduct a small RCT, including up to 50 patients and 5-15 HCPs. Eligible patients will be enrolled online. After informed consent, they will be randomized to either Pain-APP or the control group, which will consist of online educational materials (TheACPA.org). Patients in both groups will be assessed before, immediately after viewing the tool, shortly after the index clinic visit, and 1 month later. Patient-reported outcomes include patient-provider communication, pain intensity and interference, physical function, and depression (See Table 3). The investigators also include qualitative patient evaluations on a sampling (<20%) of patients to capture the full range of its impact and to explore potential mechanisms of action. Structured phone interviews, including open-ended questions, will assess patient perceptions of the platform, perceptions about how it affected communication and decisions making about treatments, trust in their HCP, and self-efficacy.

HCPs will be surveyed shortly after the patient encounter to assess acceptability of the tool, its perceived utility, and its impact on clinical efficiency. Additionally, quality of the patient encounter, ease of assessing patients with pain and of making decisions regarding treatments to manage that patient's pain will be evaluated using previously developed instruments.

The Study's Main Hypothesis: Compared to control, patients assigned to Pain-APP will have better patient-HCP communication.

Phase I data analyses plan: Multidimensional scaling was used to analyze the Nominal Group Technique (NGT) and card sort data. Hierarchical cluster analysis was used to identify subgroups of homogeneous strategies. Cognitive maps reflecting different patterns of goals and shared decision making (SDM) strategies were developed for patients and HCPs. These analyses helped the investigators understand how goals/strategies are viewed and organized by our stakeholders, which informed the design of PainApp.

Phase II data analysis plan: For the RCT, the primary outcomes analyzed will be patient-provider communication (COMM), pain (PAIN), and interference (FUNCTION), all of which will be treated as continuous.

The investigators will compare Pain-APP and the control intervention. The investigators will adhere to accepted standards. Analysis will be done in 4 stages: The investigators will examine 1) whether variables meet expected distributional assumptions; 2) bivariate associations between treatment arms and each outcome, and between covariates and outcomes; 3) unadjusted measures of effect and potential confounders; 4) exploratory multivariable analyses. Patients who are lost to follow-up will be treated according to their assigned group (intent to treat analysis). The investigators will use analysis of covariance to assess differences in outcomes between assigned groups, adjusting for any baseline differences between the randomized comparison groups. Covariates will include baseline health status, moderators listed in Table 3, and prescriber characteristics. The investigators will use linear mixed-effects models, treating scores at different points in time as repeated measures to account for inter-correlation between these measurements. The investigators will control for patient- and HCP-level factors by including them as covariates.

ii) Quantify the amount of change expected: The investigators expect to find, at minimum, a 20% improvement in communication, comparing the difference in communication pre- post- intervention in the Pain-APP group to that of the control group. Power analysis: The investigators expect a mean of 70 and a SD of 20. With the proposed sample size of 50 (25 in each arm), the investigators estimate having an 80% chance of detecting a 20% improvement on the primary outcome COMM at time=T1, with a type-I error rate of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* chronic pain for at least 1 year.
* upcoming appointment with a referring health care provider about their chronic pain within the next 3 months.

Exclusion Criteria:

* primary cause of pain due to cardiovascular or gastrointestinal problem
* unable or unwilling to give informed consent
* no access to internet
* unable to use a computer
* currently pregnant
* Unable to speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2018-06-14 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
CG CAHPS (adult, Clinician and Group Survey) | within 3 days of seeing their HCP
  The study uses a composite measure comprised of the items from the CG CAHPS survey that relate to shared decision making, including self-reported patient-provider communication (explained things, listened carefully, showed respect, spent enough time), patient rating of provider, care coordination (provider knew important information about the patient's medical history), rating of overall health and overall mental or emotional health.
The 10-item satisfaction with communication subscale of the COMRADE scale | within 3 days of seeing their HCP
  The the Combined Outcome Measure for Risk Communication and Treatment Decision Making Effectiveness (COMRADE ) (Edwards 2003) is a 20 item patient-based outcome measure, with two sub-scales for 'risk communication' and 'confidence in decision'. It is a self-reported measure of patient-provider communication. Scores from the satisfaction with communication subscale are summed to produce a total score for that subscale. A higher score corresponds to higher satisfaction. Maximum score on the subscale is 20, minimum is 0.

SECONDARY OUTCOMES:
The Brief Pain Inventory | immediately after viewing the intervention, just after seeing their HCP, and 1 month later.
  Self reported assessment of pain at its worst, least, average, and now, and interference of pain with 7 daily activities (walking, work, mood, enjoyment of life, relations with others, and sleep).
Opioid use | just after seeing their HCP and 1 month later.
  Whether or not the patient is currently using an opioid medication
The Decision Self-Efficacy Scale | immediately after viewing the intervention, just after seeing their HCP, and 1 month later.
  Self-efficacy will be measured using the Decision Self-Efficacy Scale and is a continuous variable. This scale measures self-confidence or belief in one's abilities in decision making, including shared decision making. The version with 5 response categories (0=not at all confident), 4=very confident) is used. All items are summed, divided by 11, then multiplied by 25. Scores range from 0 (not at all confident) to 100 (very confident). Higher scores (corresponding to more confidence) is considered to be better.
The Control Preference Scale | immediately after viewing the intervention, just after seeing their HCP
  The control preferences construct is defined as "the degree of control an individual wants to assume when decisions are being made about medical treatment." It is self-report, using 1-item question. These roles range from the individual making the treatment decisions, through the individual making the decisions jointly with the physician, to the physician making the decisions. Collaborative roles are generally considered preferable to the physician or patient making the decisions alone. The numerical scoring itself is not considered relevant; it is a categorical scale.
Attitude towards opioids, drawn, in part, from Prescribed Opioids Difficulty Scale | immediately after viewing the intervention, just after seeing their HCP, and 1 month later.
  Self-report of patient perception about opioids, using 1 items, intention to stop using or cut back using opioids, for people currently using an opioid. The study team adapted the question for those not using an opioid, ("It made me not want to use an opioid"; it helped me think about the pros and cons of opioids", and "It changed the way I think about opioids"

CONTACTS AND LOCATIONS:
Overall Officials: Nananda F Col, MD, Principal Investigator — Shared Decision Making Resources
Locations (1):
- Shared Decision Making Resources, Georgetown, Maine, United States

IPD SHARING:
Plan to Share IPD: Undecided
Yes, there is a plan to make individual participant data available to other researchers. It consists of a controlled access approach using a transparent and robust system to review requests and provide secure data access (reviewing all reasonable requests by our patient and clinical advisers), providing that there is adequate assurance that patient privacy and confidentiality can be maintained; and does not violate any agreements with our collaborators or sponsor organizations.

REFERENCES:
- [Background] Edwards A, Elwyn G, Hood K, Robling M, Atwell C, Holmes-Rovner M, Kinnersley P, Houston H, Russell I. The development of COMRADE--a patient-based outcome measure to evaluate the effectiveness of risk communication and treatment decision making in consultations. Patient Educ Couns. 2003 Jul;50(3):311-22. doi: 10.1016/s0738-3991(03)00055-7. PMID 12900105
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Banta-Green CJ, Von Korff M, Sullivan MD, Merrill JO, Doyle SR, Saunders K. The prescribed opioids difficulties scale: a patient-centered assessment of problems and concerns. Clin J Pain. 2010 Jul-Aug;26(6):489-97. doi: 10.1097/AJP.0b013e3181e103d9. PMID 20551723
- [Background] Sepucha KR, Borkhoff CM, Lally J, Levin CA, Matlock DD, Ng CJ, Ropka ME, Stacey D, Joseph-Williams N, Wills CE, Thomson R. Establishing the effectiveness of patient decision aids: key constructs and measurement instruments. BMC Med Inform Decis Mak. 2013;13 Suppl 2(Suppl 2):S12. doi: 10.1186/1472-6947-13-S2-S12. Epub 2013 Nov 29. PMID 24625035
- [Background] Col NF, Solomon AJ, Springmann V, Garbin CP, Ionete C, Pbert L, Alvarez E, Tierman B, Hopson A, Kutz C, Berrios Morales I, Griffin C, Phillips G, Ngo LH. Whose Preferences Matter? A Patient-Centered Approach for Eliciting Treatment Goals. Med Decis Making. 2018 Jan;38(1):44-55. doi: 10.1177/0272989X17724434. Epub 2017 Aug 14. PMID 28806143
- [Background] Degner LF, Sloan JA, Venkatesh P. The Control Preferences Scale. Can J Nurs Res. 1997 Fall;29(3):21-43. PMID 9505581
- [Derived] Col N, Hull S, Springmann V, Ngo L, Merritt E, Gold S, Sprintz M, Genova N, Nesin N, Tierman B, Sanfilippo F, Entel R, Pbert L. Improving patient-provider communication about chronic pain: development and feasibility testing of a shared decision-making tool. BMC Med Inform Decis Mak. 2020 Oct 17;20(1):267. doi: 10.1186/s12911-020-01279-8. PMID 33069228